CLINICAL TRIAL: NCT03357913
Title: Non-respiratory Comorbidities Observed in Pulmonary French Transplant Patients With Cystic Fibrosis - Exploratory Study From the French Cohort on 2004-2014.
Brief Title: Non-respiratory Comorbidities Observed in Pulmonary French Transplant Patients With Cystic Fibrosis
Acronym: MUCO TRANSPLAN
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: MUCO TRANSPLAN
Record Dates: First submitted 2017-11-20; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Pulmonary Failure; Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Lung Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Co morbidities after lung transplantation in cystic fibrosis: The population studied is the cohort of cystic fibrosis patients who received a bipulmonary transplant between 2004 and 2014 in one of the two transplantation centers in the Rhône-Alpes region.
  Interventions: Other: Lung transplantation

INTERVENTIONS:
Other: Lung transplantation — To estimate the incidence of non-respiratory co-morbidities after lung transplantation between 2004 and 2014 in the cohort of patients with cystic fibrosis grafted in the Rhône-Alpes region

SUMMARY:
Pulmonary transplantation is the reference treatment for chronic terminal respiratory failure in patients with cystic fibrosis. These are mainly bi-pulmonary transplants (cardiopulmonary transplants are exceptional). The annual number of pulmonary transplants in France for cystic fibrosis is about 90. In 2013, the transplant involves a total of more than 600 patients with cystic fibrosis. The average age at the time of the transplant is 28.5 years (2013 data, French cystic fibrosis register), compared to 58 years for patients transplanted to all pathologies. Cystic fibrosis accounts for 25% of adult bi-pulmonary grafts. Pediatric transplants are currently very rare.

The median survival after pulmonary transplantation in cystic fibrosis is currently 8.5 years (and 10 years when considering patients surviving 3 months, ie excluding early mortality). Cystic fibrosis is the pathology associated with better survival after pulmonary transplantation given the young age of patients (28.5 years on average).

The non-respiratory comorbidities associated with transplantation, all underlying pathologies combined, and referenced in the Registry of the International Society for Heart and Lung Transplantation (ISHLT) are: hypertension, diabetes, renal insufficiency, Dyslipidemia, cancers. Their frequency increases with the survival time of transplanted patients. Cystic fibrosis is associated with non-respiratory comorbidities, the frequency of which increases with age - diabetes, osteoporosis, renal insufficiency, hepatopathy, neoplastic pathologies - and may become worse after transplantation.

The main objective is to estimate the incidence of non-respiratory co-morbidities after lung transplantation in the cohort of patients with cystic fibrosis grafted in the Rhône-Alpes region.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnosis of cystic fibrosis
* Patients with Pulmonary transplant between 01/01/2004 and 31/12/2014
* Patients followed-up in one of the two pulmonary transplantation centers in the Rhône-Alpes region (Lyon, Grenoble)

Exclusion Criteria:

* Patients followed in Rhône Alpes but transplanted elsewhere in France will not be included.
* Patient refusing to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population studied is the cohort of patients with cystic fibrosis who received a bipulmonary transplant between 2004 and 2014 in one of the two transplant centers in the Rhône-Alpes region.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Incidence of co-morbidities after lung transplantation | 1 year
  The incidence rate will be calculated at 1 year follow-up after lung transplantation.
  The comorbidities studied will be:
  * diabetes
  * kidney failure
  * high blood pressure
  * hepatopathies
  * undernutrition
  * osteoporosis
  * neoplasms, and in particular colon cancer
  * gynecological complications (viral and neoplastic)
Incidence of co-morbidities after lung transplantation | 2 years
  The incidence rate will be calculated at 2 years follow-up after lung transplantation.
  The comorbidities studied will be:
  * diabetes
  * kidney failure
  * high blood pressure
  * hepatopathies
  * undernutrition
  * osteoporosis
  * neoplasms, and in particular colon cancer
  * gynecological complications (viral and neoplastic)
Incidence of co-morbidities after lung transplantation | 5 years
  The incidence rate will be calculated at 5 years follow-up after lung transplantation.
  The comorbidities studied will be:
  * diabetes
  * kidney failure
  * high blood pressure
  * hepatopathies
  * undernutrition
  * osteoporosis
  * neoplasms, and in particular colon cancer
  * gynecological complications (viral and neoplastic)
Incidence of co-morbidities after lung transplantation | 10 years
  The incidence rate will be calculated at 10 years follow-up after lung transplantation.
  The comorbidities studied will be:
  * diabetes
  * kidney failure
  * high blood pressure
  * hepatopathies
  * undernutrition
  * osteoporosis
  * neoplasms, and in particular colon cancer
  * gynecological complications (viral and neoplastic)

CONTACTS AND LOCATIONS:
Locations (1):
- Service de médecine interne Centre Hospitalier Lyon Sud, Hospices Civils de Lyon, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No